CLINICAL TRIAL: NCT06737094
Title: Prevalence and Severity of Cramps in Chronic Kidney Disease Patients
Acronym: CRAMéREIN
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240246; IDRCB-2024-A00304-43 (Other: ANSM)
Record Dates: First submitted 2024-11-28; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cramps; Chronic Kidney Disease(CKD)
Keywords: Cramps; Chronic Kidney Disease; Pain
MeSH Terms: conditions — Muscle Cramp; Renal Insufficiency, Chronic; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease (CKD) Patients: Patients with CKD stade III to V (dialysis and non dialysis)

SUMMARY:
Cramps are a frequent and severe complication in CKD patients. Their characteristics : triggering factors, associated factors, are not well known. There is no recognized effective treatment. Using a questionnaire, the investigators wish to determine prevalence, severity and associated factors of cramps in our CKD patients. Better knowledge about cramps in CKD patients will allow to better support, and give a practical tool for treatment evaluation.

DETAILED DESCRIPTION:
The investigator have elaborated a specific questionnaire for our CKD patient about cramps. This questionnaire concerns only cramps, regardless of the origin. The first question of the questionnaire will allow to evaluate the prevalence of cramps in our population of CKD patients. Every patient will indicate his medical treatment and biological datas. Only patients who will answer " Yes " to the first question will complete the cramp score of gravity questionnaire. This score is composed of 4 items : frequency of crisis, there impact on sleep, there duration and there intesity Patients will also indicate for how long time there have experimented cramps, the muscular zones involved, associated symptoms, triggering factors, and does something can help them for cramps (medicinal or non medicinal).

The third part concerns there treatment and biological datas. Finally there will complete the QOL-SF12 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary patients with CKD III to V (GFR<60ml/mn/1,72M2), including dialysed patients (hemodialysis or peritoneal dialysis).
* Non opposed to participate to the research.

Exclusion Criteria:

* Transplanted patient with functional graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient with Chronic Kidney Disease (non dialysis and dialysis patients)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cramps in CKD III-V patients. Number of patients having cramps / number of questionned patients | Day 0 - visit of inclusion

SECONDARY OUTCOMES:
Measure of Severity of cramps | Day 0 - visit of inclusion
  with a scale
Frequency of pain intensity | Day 0 - visit of inclusion
Identification of potential triggering factors | Day 0 - visit of inclusion
  through a questionnaire triggering factors will be identified
Identification of associated factors (ionic desorders, medical treatment, degree of CKD, …) | Day 0 - visit of inclusion
Identification of potential improving treatment (medicinal or not) | Day 0 - visit of inclusion
  through a questionnaire which identified potential improving treatment
Impact on Quality Of Life through a questionnaire | Day 0 - visit of inclusion
  impact of cramps on their daily life

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Alyette Costa de Beauregard, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière Service de néphrologie, Paris, France

IPD SHARING:
Plan to Share IPD: No